CLINICAL TRIAL: NCT06084689
Title: Targeting MDMD and PD1 in Tumors With Tertiary Lymphoid Structures
Acronym: EMPIRE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinuation of molecule development
Sponsor: Institut Bergonié (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2023-02; 2023-506823-28-00 (Other: EU-CTR)
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Adult Soft Tissue Sarcoma; Non Small Cell Lung Cancer; Triple Negative Breast Cancer; Colorectal Cancer; Biliary Tract Cancer
Keywords: Tertiary lymphoid structures
MeSH Terms: conditions — Sarcoma; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Biliary Tract Neoplasms; Tertiary Lymphoid Structures | interventions — brigimadlin

STUDY DESIGN:
Intervention Model Description: 2 single-arm phase II trials:
  * Cohort A: soft-tissue sarcomas
  * Cohort B: Solid tumors [non-small cell lung cancer (NSCLC) or triple negative breast cancer (TNBC) or MMS colorectal cancer (MSS-CCR) or biliary tract cancer (BTC)]
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: soft-tissue sarcomas (Experimental): Soft-tissue sarcomas
  Interventions: Drug: Ezabenlimab + BI907828
- Cohort B: Solid tumors (Experimental): Solid tumors [non-small cell lung cancer (NSCLC) or triple negative breast cancer (TNBC) or MMS colorectal cancer (MSS-CCR) or biliary tract cancer (BTC)]
  Interventions: Drug: Ezabenlimab + BI907828

INTERVENTIONS:
Drug: Ezabenlimab + BI907828 — A treatment cycle consists of 3 weeks. Both treatments will be administered on Day 1 of each cycle.

SUMMARY:
Phase II, multicenter, open-label, multi-cohort proof-of-concept study designed to evaluate the safety and efficacy of Ezabenlimab combined with BI 907828 in patients with unresectable, locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study is a phase II, multicenter, open-label, multi-cohort proof-of-concept study designed to evaluate the safety and efficacy of Ezabenlimab combined with BI 907828 in patients with unresectable, locally advanced or metastatic solid tumors.

Inclusions will proceed independently for 2 cohorts of patients with TP53 wild-type and TLS+ tumors (TLS: tertiary lymphoid strucutres), as follows:

* Cohort A: soft-tissue sarcomas

  * Single-arm phase II trial
  * 2-stage optimal Simon's design (Simon, 1989)
  * Primary endpoint: is Disease Control Rate (DCR) within 24 weeks of treatment onset, as per RECIST v1.1.
* Cohort B: Solid tumors [non-small cell lung cancer (NSCLC) or triple negative breast cancer (TNBC) or MMS colorectal cancer (MSS-CCR) or biliary tract cancer (BTC)]

  * Single-arm phase II trial
  * 2-stage optimal Simon's design (Simon, 1989)
  * Primary endpoint: is Disease Control Rate (DCR) within 24 weeks of treatment onset, as per RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis:

   * For cohort A: soft-tissue sarcoma. As recommended by the French NCI, diagnosis must be reviewed or confirmed by the RRePS Network (Réseau de référence en pathologie des sarcomes et des viscères) as recommended by the French NCI (Institut National du Cancer, Inca).
   * For cohort B: non-small cell lung cancer (NSCLC) or triple negative breast cancer (TNBC) or MMS colorectal cancer (MSS-CCR) or biliary tract cancer (BTC)
2. Age ≥ 18 years,
3. Advanced/unresectable and/or metastatic disease,
4. Mature TLS positive status
5. TP53-wild type status known (by molecular biology)
6. Cohort A: MDM2 status known at the time of inclusion
7. Cohort B: are eligible the following populations

   * NSCLC known PD-L1 tumor proportion score (TPS) < 50% AND naïve from treatment with ICI (immune checkpoint inhibitors)
   * NSCLC exposed to anti-PD1 or PD-L1 based therapy with clinical benefit (clinical benefit is defined as objective response or stable disease for at least 4 months)
   * TNBC exposed to anti-PD1 or PD-L1 based therapy with clinical benefit (clinical benefit is defined as objective response or stable disease for at least 4 months)
   * MSS-CCR naïve from treatment with ICI
   * Biliary tract cancer exposed to anti-PD1 or PD-L1 based therapy with clinical benefit (clinical benefit is defined as objective response or stable disease for at least 4 months)
8. Patients must have measurable disease (lesion in previously irradiated filed can be considered as measurable if progressive at inclusion according to RECIST v1.1) defined as per RECIST v1.1 with at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as > 10 mm with spiral CT scan.,
9. Performance status 0-2
10. Life expectancy ≥ 8 weeks,
11. Adequate hematologic and end-organ function as defined per protocol
12. Disease progression on prior treatment, or previously untreated disease with no available acceptable treatment
13. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment (excluding alopecia and vitiligo of any grade and non-painful peripheral neuropathy grade ≤ 2) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 5.0),
14. Ability to comply with the study protocol, in the investigator's judgment
15. Female subjects of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study treatment. Serum or urine pregnancy test must be repeated within 72 hours prior to receiving the first dose of study medication,
16. Both women of childbearing potential and men must agree to use two medically acceptable methods of contraception throughout the treatment period
17. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for: a. superficial/non-invasive bladder cancer, or basal or squamous cell carcinoma in situ treated with curative intent; b. endoscopically resected GI cancers limited to the mucosal layer without recurrence in > 1 year,
18. Voluntarily signed and dated written informed consent prior to any study specific procedure,
19. Patients with a social security in compliance with the French law.

Exclusion Criteria:

1. Prior treatment with ezabenlimab and/or BI 907828,
2. Women who are pregnant or breast feeding,
3. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
4. Previous enrolment in the present study,
5. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons,
6. Inability to swallow,
7. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins,
8. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the ezabenlimab or BI 907828 formulation,
9. Symptomatic or actively progressing central nervous system (CNS) metastases.
10. History of leptomeningeal disease,
11. Primary CNS tumors with any of the following characteristics:

    * History of intracranial hemorrhage or spinal cord hemorrhage
    * Neurosurgical resection or brain biopsy to the primary brain tumor within 28 days of Cycle 1 Day 1
12. Any systemic anticancer treatment within 2 weeks or 5 half-lives (whichever is shorter) prior to start of ezabenlimab combined with BI 907828,
13. Whole brain radiotherapy within 14 days prior to start of BI 754091 combined with BI 907828
14. Stereotactic radiosurgery within 7 days prior to start of ezabenlimab combined with BI 907828
15. Active bleeding, significant risk of haemorrhage (e.g. previous severe gastrointestinal bleeding, previous haemorrhagic stroke at any time), or current bleeding disorder (e.g. haemophilia, von Willebrand disease)
16. History of or concurrent serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study or confounds the ability to interpret data from the study
17. Incomplete recovery from any surgery prior to the start of ezabenlimab combined with BI 907828 that would interfere with the determination of safety or efficacy of ezabenlimab combined with BI 907828
18. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or higher), myocardial infarction, or cerebrovascular accident within 3 months prior to enrollment, unstable arrhythmias, or unstable angina
19. Uncontrolled tumor-related pain.
20. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
21. Active or history of autoimmune disease or immune deficiency,
22. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
23. Active tuberculosis
24. Severe infection within 4 weeks prior to initiation of ezabenlimab combined with BI 907828, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
25. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of ezabenlimab combined with BI 907828.
26. Prior allogeneic stem cell or solid organ transplantation
27. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of ezabenlimab combined with BI 907828, or anticipation of need for such a vaccine during treatment or within 6 months after the final dose ezabenlimab combined with BI 907828. Seasonal flu vaccines that do not contain a live virus are permitted,
28. Current treatment with anti-viral therapy for HBV
29. Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to initiation of ezabenlimab combined with BI 907828
30. Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of ezabenlimab combined with BI 907828, or anticipation of need for systemic immunosuppressive medication during ezabenlimab combined with BI 907828.
31. Patients with oral anticoagulation based on Vitamin K antagonist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 6 months
  Disease control rate (DCR), defined as the proportion of patients with disease control lasting for at least 24 weeks since treatment onset, will be reported.

SECONDARY OUTCOMES:
Objective response rate | 6 months
  Objective response rate (ORR), defined as the proportion of patients with objective response will be assessed, based on centralized radiological review, within 24 weeks of treatment onset.
Duration of response (DoR) | 1 year
  Duration of response (DoR) defined as the time from documentation of tumor response (CR, Cru, PR, PRu) to disease progression (as per RECIST V1.1).
Progression-free survival (PFS) | 1 year
  Progression-free survival (PFS) defined as the time from the first day of treatment to the first documented disease progression (as per RECIST v1.1) or death (due to any cause), whichever occurs first.
Overall survival | 1 year
  Overall survival defined as the time from the first day of treatment to death (due to any cause).
Safety and tolerability of the combination | Throughout treatment period, an expected average of 6 months
  Occurence of adverse events (AEs) and Serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ITALIANO, MD, PhD, Principal Investigator — Institut Bergonié
Locations (6):
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHRU Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes